CLINICAL TRIAL: NCT07319260
Title: All Children Underwent Congenital Heart Disease (CHD) Surgery Under General Anesthesia. The Intervention Group and Control Group Each Had 35 Children. The Control Group Received Routine Pain Care, While the Intervention Group Received Nursing Based on Animated Film-based Nurse-patient Interactive Mode in Addition to Routine Pain Care.
Brief Title: Application of Nurse-Patient Interaction Model Based on Animated Cartoons in Postoperative Analgesia for Preschool Children With Congenital Heart Disease.
Acronym: CCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BeijingChildrens xinwai; ［2024］-Y-199-D (Other: Capital Medical University Affiliated Beijing Children's Hospital)
Record Dates: First submitted 2025-12-09; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: A Study on the Effect of Animation-based Nurse-Patient Interaction Model on Postoperative Pain in Children With Congenital Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Based on the nurse-patient interaction model in animated cartoons (Experimental): Establish an animation database: Since children of different ages prefer different cartoons, and considering that each child has different individual psychological characteristics, each child likes different cartoons. When using cartoons, to ensure that the cartoons have a certain level of appeal to the children and capture each child's attention, the research team established an animation database before the intervention group was implemented. This allows nursing staff to watch and select the 3 favorite cartoons with the child before the procedure.They were cared for by the same group of nursing staff as the control group, but before the intervention, during the interval period, the researchers completed training on the implementation plan of the patient-nurse interaction model based on animated films and the data collection methods for the intervention group.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Routine care — Routine care
  Other Names: Control group Routine postoperative care

SUMMARY:
I. Research Objective To verify the efficacy of an animated nurse-patient interaction model in alleviating postoperative pain in children with congenital heart disease, optimize non-pharmacological analgesic nursing processes for children post-surgery, and improve family nursing satisfaction.

II. Research Subjects Thirty-five children aged 3-7 years who underwent curative surgery for congenital heart disease were selected and randomly divided into an observation group and a control group, each consisting of 35 cases.

* Inclusion criteria: Normal cognitive function, admitted to the intensive care unit post-surgery, and family informed consent obtained.
* Exclusion criteria: Concurrent severe organ or neurological diseases, occurrence of severe postoperative complications, or resistance to animated intervention.

III. Research Methods

1. Intervention Measures

   * Control group: Implemented routine postoperative pain management for congenital heart disease (pharmacological analgesia + basic nursing).
   * Observation group: On the basis of routine nursing, preoperative assessment of children's animated preferences was conducted. Appropriate-age animations were played 15-30 minutes per session, 3-4 times per day when the child's vital signs were stable post-surgery. Nurses synchronized interactive activities, and pain was assessed every 2 hours, with intervention strategies adjusted based on scoring.
2. Observation Index

   - Secondary indicators: Child anxiety score, family anxiety score (SAS), nursing satisfaction.
3. Statistical Analysis: SPSS 26.0 software was used. t-test was performed for measurement data, and χ² test was performed for counting data. P < 0.05 was considered as statistically significant difference.

IV. Implementation Steps 1. Preparation Phase: Form a team, develop the protocol and informed consent form, and train the researchers. 2. Intervention phase: Recruitment and grouping of subjects, implementation of interventions, and data collection. 3. Analysis and Summary Phase: Conduct statistical analysis of data, prepare reports, and establish standardized nursing procedures.

V. Ethics and Expected Outcomes Ethics: With approval from the hospital's ethics committee and after obtaining informed consent from the family, the child may voluntarily withdraw from the study. The control group will receive equivalent intervention opportunities after completing the study.

DETAILED DESCRIPTION:
Research Protocol for Postoperative Pain Management in Children with Congenital Heart Disease Based on the Animation-Patient Interaction Model Background and Objectives (1) Research Background Congenital heart disease is one of the common congenital malformations in children, with surgical intervention being the primary treatment modality. Postoperative wound pain and catheter irritation can easily trigger crying and agitation in pediatric patients, not only impairing wound healing and postoperative recovery but also increasing psychological burden on parents. Traditional pain management primarily relies on pharmacological analgesia, which carries certain side effects. Moreover, young patients exhibit limited capacity for pain expression, making precise assessment and intervention challenging. The animation-patient interaction model represents an innovative approach that integrates age-appropriate animated content into perioperative care. By diverting children's attention and alleviating negative emotions, this method reduces pain perception, providing a novel non-pharmacological intervention direction for postoperative pain management in pediatric patients.

(2) Research Objectives 1. To evaluate the efficacy of the animated nurse-patient interaction model in improving postoperative pain scores, crying duration, and sleep quality in children with congenital heart disease.

2. To explore the impact of this model on anxiety levels and nursing satisfaction among family members of pediatric patients.

3. Develop a standardized and scalable animated nursing process for postoperative patient-nurse interaction in children with congenital heart disease.

2. Study Subjects and Methods (1) Study Subjects The study subjects were children undergoing radical surgery for congenital heart disease in the Department of Cardiac Surgery of a tertiary Grade A children's hospital. The inclusion and exclusion criteria were as follows: 1. Inclusion Criteria-Age 3-7 years, with normal cognitive function and the ability to normally watch animations; -Scheduled for elective radical surgery for congenital heart disease, requiring postoperative admission to the intensive care unit (ICU) for observation; -Informed consent from the child's family members, with voluntary participation in the study.

2. Exclusion criteria: -Concomitant severe organ diseases or neurological disorders; -Postoperative severe complications (e.g., massive hemorrhage, septic shock, etc.); -Significant emotional resistance to the animated content.

A controlled trial was conducted, with eligible pediatric patients divided into an observation group and a control group at a 1:1 ratio, each comprising 35 cases. (II) Research Methods 1. Intervention Method-Control Group: The conventional postoperative pain management protocol for congenital heart disease was implemented, including prescribed analgesics, positional care, wound care, and basic psychological reassurance.

* Observation Group: In addition to conventional pain management, the animation-based nurse-patient interaction model was implemented, with the specific intervention process as follows: ① Preoperative assessment: The nurse evaluated the child's age and interest preferences one day before the procedure, communicated with the family to determine the type of animation the child preferred, and selected age-appropriate animations that were non-violent, slow-paced, and visually soothing (e.g., Peppa Pig, Super Wings, etc.), while preparing mobile playback devices.

  * Postoperative intervention: After the child regains consciousness and stabilizes vital signs postoperatively, selected animations are played in the intensive care unit (ICU) for 15-30 minutes each session, 3-4 times daily. During playback, nurses conduct synchronous nurse-patient interaction, such as explaining the animation plot and guiding the child to imitate the actions of the animated characters. Concurrently, the FLACC pain scale is used to assess the child's pain level every 2 hours.

    * Intervention adjustment: Optimize the intervention strategy based on pain scores. For mild pain, focus on animation playback and interaction; for moderate pain, combine non-pharmacological nursing measures such as massage and position adjustment; for severe pain, supplement with animation intervention in addition to prescribed medication.

      2. Observation indicators-Primary indicators: Pain scores of pediatric patients at 1 hour, 6 hours post extubation, and 24/48 hours postoperatively.

Secondary indicators: anxiety scores of pediatric patients, anxiety scores of family members (using the Self-Rating Anxiety Scale, SAS); nursing satisfaction scores (using a hospital-developed nursing satisfaction questionnaire).

3. Data Collection and Statistical Analysis-Trained researchers were assigned to collect data, ensuring its objectivity and accuracy.

-Data analysis was performed using SPSS 26.0 statistical software. Measurement data were expressed as mean ± standard deviation, and intergroup comparisons were conducted using t-test. Categorical data were expressed as rates, and intergroup comparisons were performed using χ² test. A P-value <0.05 was considered statistically significant.

III. Research Content and Implementation Steps (1) Research Content 1. Standardization process construction of the animated patient-nurse interaction model, including animation screening criteria, playback timing, interaction methods, and effect evaluation dimensions.

2. Comparative analysis of postoperative pain-related indicators and rehabilitation indicators between the observation group and the control group.

3. Investigation and analysis of the psychological status and nursing satisfaction of pediatric patients' family members.

(2) Implementation Steps 1. Preparation Phase: Establish a research team comprising cardiac surgery nurses, pediatric nursing researchers, and statistical analysts; develop the research protocol and informed consent form; train researchers to standardize intervention methods and data collection criteria.

2. Intervention phase: Recruit study subjects, randomly assign them to groups, and implement corresponding interventions; strictly collect all index data according to the study protocol, and promptly record and organize the data.

3. Data analysis phase: Input and statistical analysis of collected data, comparison of index differences between the two groups, and verification of intervention efficacy.

4. Summary phase: Prepare the research report, establish standardized nursing procedures, and propose recommendations for clinical implementation.

IV. Ethical Considerations 1. This research protocol was implemented after approval by the hospital ethics committee.

2. Before the study, provide detailed explanations to the child's family regarding the purpose, methods, risks, and benefits of the study, and obtain their informed consent. During the study, respect the child's wishes, and allow them to withdraw from the study at any time if they exhibit resistance.

3. The control group received conventional nursing care, and after the study concluded, equal opportunities for animated care-intervention interactions were provided to the children in the control group to safeguard their rights.

V. Promotional Value This model is characterized by its simplicity, low cost, and high safety, making it suitable for widespread application in pediatric and cardiac surgery departments across all levels of hospitals. It not only enhances the quality of postoperative pain management in children but also optimizes the nurse-patient relationship and improves family satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Children diagnosed with CHD and treated with surgical intervention according to the 'Pediatric Congenital Heart Disease Diagnosis and Treatment Guidelines' and echocardiographic images [100];

    * Age between 3 to 7 years, including 3 years and 7 years;

      * Surgical procedure is thoracotomy;

        * Diagnosed with ventricular septal defect, atrial septal defect, or atrial septal defect combined with ventricular septal defect, patent ductus arteriosus, or tetralogy of Fallot;

Exclusion Criteria:

* Inclusion criteria:

  * Children diagnosed with CHD and treated with surgical intervention according to the 'Pediatric Congenital Heart Disease Diagnosis and Treatment Guidelines' and echocardiographic images [100];

    * Age between 3 to 7 years, including 3 years and 7 years;

      * Surgical procedure is thoracotomy;

        ④ Diagnosed with ventricular septal defect, atrial septal defect, or atrial septal defect combined with ventricular septal defect, patent ductus arteriosus, or tetralogy of Fallot;

Ages: 3 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-08-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Assessment in Children with Congenital Heart Disease | 1 hours after tube removal to 48 hours after surgery
  Pain scores at 1 hour, 6 hours, 24 hours, and 48 hours after extubation
Pain Assessment | The responsible nurse used the Wong-Baker Facial Expression Scale to assess pain at 1 hour, 6 hours after tube removal, 24 hours, and 48 hours post-operation, and recorded the scores on the corresponding assessment forms. The researchers reviewed these a
  This study used the Wong-Baker FACES Pain Rating Scale for pain assessment in children. The Wong-Baker FACES Pain Rating Scale was originally developed by Donna Wong and Dr. Connie Baker for measuring children's pain. It was later revised to form the FPS-R scale. This method began to be used in clinical assessment in 1990. It uses six facial expressions ranging from smiling to crying to represent different degrees of pain. During assessment, the child only needs to select one expression that represents their pain level (see Figure 1 for details). The total score is 10 points, where 0-3 indicates no pain or mild pain; 4-7 indicates moderate pain; and 8-10 indicates severe pain. This scale has a wide range of applications, suitable for children of all ages, does not require the child to have a specific cultural background, and is easy to master. Studies by Garra et al.have validated the effectiveness of the Wong-Baker FACES Pain Rating Scale. Studies by Newman et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Study on the effect of cartoon nurse-patient interaction mode on postoperative pain in children with congenital heart disease, Beijing, China

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT07319260/Prot_SAP_ICF_000.pdf